CLINICAL TRIAL: NCT01176695
Title: A Randomized, Double Blind, Controlled, Parallel Group, Multicenter Study on the Efficacy and Safety of a Fish Oil Containing Lipid Emulsion vs. a Medium and Long Chain Lipid Emulsion in Patients Undergoing Elective Abdominal Surgery of Moderate Severity
Brief Title: Efficacy and Safety of a Fish Oil Containing Lipid Emulsion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-0802
Record Dates: First submitted 2010-05-10; First posted 2010-08-06 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): fish oil containing lipid emulsion
  Interventions: Drug: fish oil containing lipid emulsion
- 2 (Active Comparator): MCT/LCT containing lipid emulsion
  Interventions: Drug: MCT/LCT containing lipid emulsion

INTERVENTIONS:
Drug: fish oil containing lipid emulsion — medium chain triglycerides, long chain triglycerides, omega-3 fatty acid containing triglycerides
  Arms: 1
Drug: MCT/LCT containing lipid emulsion — medium chain triglycerides, long chain triglycerides
  Arms: 2

SUMMARY:
The purpose of the study is to compare a fish oil containing lipid emulsion against a medium-chain/long-chain triglyceride (MCT/LCT) lipid emulsion in terms of their efficacy and safety during postoperative parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patients considered for open abdominal surgery of moderate severity, e.g.. radical operation for stomach cancer or pancreaticoduodenal surgery
* Male and female patients ≥18 and <85 years of age
* Indication for total parenteral nutrition therapy: for at least 5 consecutive days after operation
* Ability and willingness to give voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Institutional Review Board (IRB) prior to all evaluations, and to comply with the requirements of the study.

Exclusion Criteria:

* General contraindications for parenteral nutrition (acidosis of various geneses, untreated disorders of electrolyte and fluid intake and output, inadequate cellular oxygen supply)
* General contraindications for infusion therapy such as acute pulmonary oedema, hyperhydration and decompensated cardiac insufficiency
* Known hypersensitivity to egg-, soy-, and fish proteins or any of the ingredients
* Other

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To investigate on the efficacy of fish oil on the nutrition status | day 1 to day 6
  Prealbumin as the primary endpoint variable
To investigate on the efficacy of fish oil on an inflammatory parameter | day 1 to day 6
  LTB5/LTB4 as a second primary endpoint

SECONDARY OUTCOMES:
Incidence of postoperative complications | 6 days
Liver function | 6 days
Coagulation parameters | 6 days
Blood chemistry | 6 days
SIRS | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Prof. MD. PhD., Principal Investigator — Nanjing Hospital
Locations (2):
- China (2):
  - Hospitals, Beijing
  - Nanjing Hospital, Nanjing